CLINICAL TRIAL: NCT00055354
Title: Acupuncture Diagnosis and Treatment of DSM-IV PTSD
Brief Title: Acupuncture for the Treatment of Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT001229-01 (NIH)
Record Dates: First submitted 2003-02-26; First posted 2003-02-27 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Acupuncture; Medicine, Chinese Traditional
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Acupuncture Therapy; Cognitive Behavioral Therapy

INTERVENTIONS:
Procedure: Acupuncture
Behavioral: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to evaluate acupuncture as a treatment for Post-Traumatic Stress Disorder (PTSD) and to correlate the diagnosis of PTSD with Traditional Chinese Medicine (TCM) diagnostic patterns.

DETAILED DESCRIPTION:
This study will evaluate: 1) the TCM diagnostic differentiation patterns of people who have PTSD as defined by the Diagnostic and Statistical Manual, 4th edition; 2) if an acupuncture treatment approach is acceptable to people with PTSD; and 3) if an acupuncture treatment approach is associated with a reduction in PTSD symptoms that is comparable to that of standard treatments. Because symptoms of depression, insomnia, and pain are often associated with PTSD, we will also evaluate the potential benefit of an acupuncture approach to depression, insomnia, and pain symptoms in people with PTSD.

Patients in this study will be randomized to one of three groups. Group A will receive acupuncture therapy. Group B will receive standard Cognitive Behavior Therapy. Group C is a control group and will receive no treatment. Patients in Groups A and B will undergo a total of 24 hours of therapy over the 3 month study course. All patients will have five nontherapeutic study visits; these visits will address diagnosis and assessment. Study visits will include assessments of PTSD symptoms, sleep symptoms, and level of impairment.

ELIGIBILITY:
Inclusion Criteria

* DSM-IV diagnosis of PTSD
* Stage I PTSD symptoms
* PTSD Symptom Scale-Self Report (PSS-SR) score > 16
* Meets PSS-SR diagnostic criteria

Exclusion Criteria

* Stage I substance abuse and/or dependence in the past 6 months
* Psychotic disorder
* Inability to commit to treatment or wait-list conditions
* Current treatment specifically for PTSD
* Certain medical conditions, including thyroid disease, class IV heart failure, active cancer treatment, and uncontrolled diabetes
* Pregnant
* Use of benzodiazepines, narcotics, opiates, narcotic antagonists, sleep medication, muscle relaxants, analgesics, or sedatives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2002-09; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Health Sciences Center- Department of Psychiatry, Albuquerque, New Mexico, United States